CLINICAL TRIAL: NCT03866616
Title: Evaluation Study of the Impact of the New Brain Builders Parenting Class Offered at WIC Clinics
Brief Title: Evaluation Study of the Impact of the New Brain Builders Parenting Class
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The PI discontinued the evaluation study.
Sponsor: William Marsh Rice University (Other)
Collaborators: Harris County Department of Public Health (Unknown); City of Houston Department of Health and Human Services WIC offices (Unknown); Episcopal Health Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-216
Record Dates: First submitted 2019-02-11; First posted 2019-03-07 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Child Development; Mother-Child Interaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (usual care) (Active Comparator): Behavioral: This arm receives usual care ("control group") consisting in: WIC participants will attend their usual appointments completed at the WIC clinics.
  Interventions: Behavioral: Control (Usual care)
- Intervention (group sessions) (Experimental): Behavioral: Brain Builders Parenting Class-intervention (BBPC). Participants who are selected via the lottery to participate in the BBPC program will be asked to attend six, 1-hour classes, every other week over a 12 week period of time.
  Interventions: Behavioral: Brain Builders Parenting Class

INTERVENTIONS:
Behavioral: Brain Builders Parenting Class — Brain Builders Parenting Class group sessions goal is to increase parental knowledge of brain development and increase responsive parenting
  Arms: Intervention (group sessions)
Behavioral: Control (Usual care) — This arm receives usual care ("control group") consisting in: WIC participants will attend their usual appointments completed at the WIC clinics.
  Arms: Control (usual care)

SUMMARY:
The objective of this research is to evaluate the effectiveness of the parenting program on increasing positive parent-child interactions and increasing cognitive achievement in children. Overall, this project is intended to benefit women and children and supplement WIC services.

The Brain Builders Parenting Class Evaluation Study Research Questions include the following:

1. Does the program impact child development outcomes such as kindergarten readiness?
2. Does the program increase parental knowledge about the importance of high-quality parent-child interaction for child development?
3. Does the program impact the quality and quantity of the parent-child interactions?

DETAILED DESCRIPTION:
Science demonstrates that the foundation of a person's ability to be innovative, creative, analytical and intellectual is established in the brain during the first few years of life. The brain controls every aspect of human life, from breathing to learning, behaving, adapting and thinking. Because the brain controls all aspects of human life, impaired brain function compromises physical, mental, and emotional health and overall productivity in society. The parent-child or caregiver-child relationship is one of the most important experiences for brain development and cognitive outcomes in young children. This relationship is vital for optimal brain development because of the dependency of neuronal connections on stimulating human interaction. Parental response to their child's verbal or nonverbal cues, frequently called "serve and return", influences whether neural connections are strengthened or eliminated. An example of a positive serve and return scenario is a caregiver or parent's attentive response to a young child's cries through eye contact, acknowledging the child, and meeting the child's need. This type of positive interaction fosters neural connections that are important for communication and social skills.

Many parents do not know or understand the impact their responses have on their child's brain development. While there are many parenting programs that teach parenting skills and behaviors, there were no evidences of any programs that were culturally and economically sensitive to vulnerable families and also educated parents on the brain science as well as equip parents with the skills to be responsive parents Brain Builders Parenting Class will work with both inner city and rural WIC clinics with representative populations of pregnant women and women with children under 1 years old, to provide parenting programs, led by WIC staff focused on brain development.

The study will evaluate the effectiveness of the parenting program in increasing positive parent-child interactions and increasing cognitive achievement in the children. The main goal of this evaluation study is to increase parents' self-efficacy by increasing their knowledge of brain development, improve their skills through observational learning and behavioral capability, provide reinforcement for positive interactions with baby and child, and increase their social support through the group parenting classes and shared experiences. The evaluation study will have two rounds. The first round will take place at recruitment in the WIC Centers. The second round will take place around the time that the child is between 22 and 26 months old. This visit will take place at the WIC clinic.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking healthy women who have not had a prior live birth and are between their 13th and 22nd week of pregnancy, English-speaking healthy women who are between their 13th and 22nd week of pregnancy and and who have children 6 years or older;
* English-speaking healthy women: First time mothers of 0 to 1-year old children
* English-speaking healthy women: Mothers of 0 to 1-year old children who have children 6 years or older;
* Are at least 18 years old, AND (2) self-identify as non-Hispanic white, Hispanic/Latinx, Asian or black/African American
* Are not planning to move to a location more than 50 miles from the WIC clinic in the first two years after the baby's birth;
* Are not planning to put the baby up for adoption
* Women who agreed to participate in the lottery for the Brain Builder Parenting Class program.
* Women who are pregnant with multiples (i.e. twins, triples, etc) will also be eligible for participation.
* Children of healthy women who are enrolled in the pilot evaluation study
* Children between the ages of 0-12 months at the time of recruitment. -

Exclusion criteria:

* Non-English-speaking women;
* The woman is not between her 13th and 22nd week of pregnancy
* The woman has more than one biological child
* The woman does not participate in the WIC clinic
* The woman is planning to move to a location more than 50 miles from WIC clinic in the two years after the baby's birth;
* The woman is planning to put the baby up for adoption;
* The woman does not agree to participate in the lottery for the Brain Builder Parenting Class program.
* English-speaking healthy women:
* First time mothers of 0 to 1-year old children
* Children of healthy women who are not enrolled in the pilot evaluation study. Children that are not between the ages of 0-12 months at the time of recruitment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2019-06-24 (Actual); Primary Completion 2019-12-15 (Actual); Study Completion 2019-12-15 (Actual)

PRIMARY OUTCOMES:
Child Development | Measured at 22 to 26 months of age
  The child development will be assessed by using the Caregiver Reported Early Development Index (CREDI). The CREDI measures five dimension of child development: Motor development, Language development; Socioemotional development; Cognitive development; and Mental health. The CREDI was designed to serve as a population-level measure of early childhood development for children from birth to age three. As the name suggests, the CREDI exclusively relies on caregiver reports, and thus primarily focuses on milestones and behaviors that are easy for caregivers to understand, observe and describe.
Quality of the Language Environment: LENA System | Measured at 22 to 26 months of age
  The quality of the language environment at home will be measured by using the LENA System (LENA). LENA is an integrated processing and cloud-based software package that enables researchers to collect, manage, and analyze multiple recordings of children ages 2 months to 48 months.LENA device estimates adult words spoken to and around the key child, adult-child conversational interactions, child vocalizations, and language from TV and/or electronics
Measurement of the Child's Home Environment | Measured at 22 to 26 months of age
  The StimQ instrument is a 39-point scale for measuring cognitive stimulation in the homes of children. It includes four sub scales: Availability of Learning Materials (ALM); Reading Scale; Parental Involvement in the Developmental Advance (PIDA); and Parental Verbal Responsivity (PVR). The ALM describes the type of learning materials available to a child. The Read Scale measures the number of books in the home and the amount of days spent reading to the child. The PIDA is scored by the number of 'Yes' responses to ten questions regarding parental involvement in child development. The PVR is scored by calculating the total number of 'Yes' responses to four questions regarding parental verbal responsibility. Higher values are associated with a better outcome since a higher value indicates the presence of more learning materials in the home. Subscales are combined by summing all the subscale scores to get the total StimQ score.
Parenting Interactions with Children: Checklist of Observations Linked to Outcomes (PICCOLO). | Measured 22 to 26 months of age
  This scale measures the presence and absence of 29 developmentally supportive parenting behaviors across the entirety of a 10 minute, video recorded interaction. The PICCOLO scale is divided into four subcategories: affection, responsiveness, encouragement, and teaching. Each subcategory has approximately 7-8 parenting behaviors that a PICCOLO practitioner would observe. Each category's behaviors are scored on a scale from 0-2 where parents receive (0) if none of the behavior, (1) if some of the behavior, (2) if lots of the behavior. Higher values are associated with better outcomes since high values indicate a high amount of affection, responsiveness, encouragement, and teaching, which are behaviors linked to healthy cognitive development in children
Quality of the Child Sleep: The Brief Infant Sleep Questionnaire (BISQ) | Measured at 22 to 26 months of age
  The Brief Infant Sleep Questionnaire (BISQ) was developed on the basis of a review of the infant sleep literature in search of meaningful variables, particularly clinical studies based on the use of subjective and objective infant sleep measures. The questionnaire variables included 1) nocturnal sleep duration; 2) daytime sleep duration); 3) number of night wakings; 4) duration of wakefulness during the night hours; and 5) nocturnal sleep-onset. The criteria used to define poor sleepers on the basis of the BISQ measures are as follows: 1) the child wakes > 3 times per night; 2) nocturnal wakefulness period is > 1 hour; or 3) the total sleep time is < 9 hours. Soothing techniques and the location of sleep are also evaluated and seem to play important roles in infant sleep. Infants who fall asleep alone in the crib and sleep in a crib in a separate room are more likely to sleep through the night, with fewer night wakings
Parent's beliefs | Measured at baseline and from 22 to 26 months of age
  The parent's beliefs questionnaire measures the impact of parental investments in the child (for example, reading to the child) on child development.

SECONDARY OUTCOMES:
Center for Epidemiological Studies Depression Scale (CES-D) | Measured at baseline
  Maternal depressive symptomatology measured by the Center for Epidemiological Studies Depression Scale (CES-D)The score is the sum of the 20 questions. Each question has a total of four responses to choose from and each response is scored from 0-3 respectively.Possible range is 0-60. A score of 16 points or more is considered depressed. High values are considered a worse outcome since a score of 16 points or higher is indicative of depression.

CONTACTS AND LOCATIONS:
Overall Officials: Snejana Nihtianova, PhD, Principal Investigator — William Marsh Rice University
Locations (2):
- United States (2):
  - Northeast WIC Center, Houston, Texas
  - Harris County Public Health Antoine WIC, Houston, Texas